CLINICAL TRIAL: NCT06611111
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled Trial of Pulse Dosed Ceftriaxone for Post-Treatment Lyme Disease
Brief Title: Ceftriaxone Pulse Dose for Post-Treatment Lyme Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-02-UMU
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-02

CONDITIONS: Post-Treatment Lyme Disease
Keywords: Pulse Dose; Ceftriaxone; PTLDS; Chronic Lyme Disease
MeSH Terms: conditions — Post-Lyme Disease Syndrome | interventions — Ceftriaxone; Glucose

STUDY DESIGN:
Intervention Model Description: Participants who meet inclusion/exclusion criteria will be randomized 1:1 into receiving ceftriaxone or placebo. At day 181, the study will be unblinded and participants in the placebo group will be invited to receive ceftriaxone on the same schedule.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ceftriaxone (Active Comparator): Participants will receive IV infusion of 2g Ceftriaxone, approximately every 5 days for 6 weeks for a total of 9 treatments.
  Interventions: Drug: Ceftriaxone (Rocephin®)
- Placebo (Placebo Comparator): Participants will receive IV infusion of dextrose 5% in water, approximately every 5 days for 6 weeks for a total of 9 treatments
  Interventions: Drug: Dextrose 5% (D5W)

INTERVENTIONS:
Drug: Ceftriaxone (Rocephin®) — Slightly yellow liquid.
  Arms: Ceftriaxone
Drug: Dextrose 5% (D5W) — Colorless liquid
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if an FDA approved drug, Ceftriaxone, given intermittently, can treat people between 18 and 75 years old with a history of Lyme disease, who are still experiencing persistent or returning symptoms after they have completed treatment. The main questions it aims to answer are:

* Will giving Ceftriaxone approximately every 5 days for 6 weeks be safe and well tolerated when compared to a group that receives placebo (a look-alike substance that contains no drug)?
* Will giving Ceftriaxone improve symptoms?

Participants will be asked to do the following:

* Come to the clinic approximately every 5-6 days to receive an IV infusion of either the Ceftriaxone or placebo.
* Answer questions about their level of tiredness, body pain, general health and physical ability, sleep, anxiety, depression and any suicidal thoughts.
* Give blood so we can make sure your body is handling the drug okay or to help us learn more about how the drug is affecting the persistent Lyme disease symptoms.

DETAILED DESCRIPTION:
This study will explore treating participants who are 18 to 75 years old with Post-Treatment Lyme Disease. IV Ceftriaxone will be delivered in a pulse dose fashion, approximately every 5 days for a total of 9 IV infusions over 6 weeks. Participants will return one month following last treatment, at approximately 3 and 6 months from study start. At each study visit, participants will be asked a number of questionnaires including the SAFTEE assessment to assess the side effects of the drug as compared to placebo; the Fatigue Severity Scale, SF-36, GSQ-30, and PROMIS-29 questionnaires to assess physical functioning, general health, vitality, social functioning, bodily pain, role physical, role emotional, mental health, symptoms, fatigue, anxiety, depression, and sleep disturbances; the CSSRS to assess suicidal ideation.

At the 6-month mark, the study will be unblinded and participants in the placebo group will be invited to repeat the study visits receiving Ceftriaxone. Participants who originally received Ceftriaxone will receive a phone call follow up at 1 year. The duration for both groups is one year. Samples will be collected for safety labs and research assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 at the time of consent
2. Ability and willingness to sign informed consent
3. Available for the study period
4. Must have met the definition of a prior well-defined or probable Lyme disease infection, AND meet the definition of PTLDS
5. Provide consent for release of medical history records from primary care physician, college or university, urgent care or emergency room visit
6. Have a level of fatigue that interferes with their ability to function in their job, schooling, or other social/personal activities (FSS score of 4 or higher)
7. Subjects will need to have been off of antibiotics (those standard antibiotics used to target Lyme disease to include doxycycline, amoxicillin, cefuroxime, azithromycin, ceftriaxone or penicillin) for at least 6 weeks prior to study enrollment and be willing to remain off of any outside antibiotics during the duration of the treatment component of the study.

Exclusion Criteria:

1. Female: pregnant or lactating
2. Women who intend to become pregnant during the treatment study period (approximately 45 days)
3. Patients with a diagnosis of Lyme disease based on only a positive Lyme IgM immunoblot
4. A history of cephalosporin allergy or significant intolerance
5. Lyme related symptoms that have been present for greater than 10 years
6. Blood tests confirming infection with human immunodeficiency virus- 1 (HIV-1), hepatitis C, hepatitis B (assessed by HbsAg) virus.

   Note: Subjects who have well controlled HIV, who are on ART with a CD4 count greater than 200 will be allowed to participate.
7. Diagnosis with Bipolar Disorder or Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition (to include any finding of increased suicide risk as identified by a rating of moderate or high risk on the CSSRS assessment), which in the opinion of the investigator prevents the subject from participating in the study
8. Known concurrent rheumatologic or similar disease thought to interfere with study participation or confound results at the discretion of the investigator. These may include but are not limited to rheumatoid arthritis, systemic lupus erythematous, Sjogren's syndrome, scleroderma, psoriasis, fibromyalgia, chronic fatigue syndrome/myalgic encephalomyelitis, or obstructive sleep apnea
9. Hives, shortness of breath, swelling of the lips or throat, or hospitalization related to a previous treatment with a cephalosporin antibiotic, or severe allergic reaction to penicillins (e.g. anaphylaxis or severe rash with Stevens Johnson syndrome or similar)
10. Planned travel during the study period that would interfere with the ability to complete all study visits (this can be a temporary exclusion with plan to schedule enrollment during a window of time during which they could attend their study visits)
11. Significant screening physical examination abnormalities or chronic medical condition that in the opinion of the investigator may impact subject safety
12. 12. Participation (active or follow-up phase) or planned participation in another vaccine, drug, or medical device in the 4 weeks prior to this trial, within 5 times the elimination half-life, whichever is longer, or during the trial
13. Prior history of Clostridium difficile infection
14. Currently taking warfarin (Coumadin)
15. Unable to comply with study requirements
16. Clinician discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of abnormal laboratory measurements | 30 days post last treatment
  Total number of all abnormal labs
Intensity of Abnormal Laboratory Measurements | 30 days post final treatment
  Graded according clinical laboratory normals and FDA toxicity scale
Duration of Abnormal Laboratory Measurements | 30 days post final treatment
  Number of days of abnormal lab
Occurrence of adverse events | 30 days post last treatment
  Total number of adverse events
Intensity adverse events | 30 days post final treatment
  Graded according FDA toxicity scale
Duration of adverse events | 30 days post final treatment
  Number of days per adverse event
Number of serious adverse events | 1 year post study start
  Total number

SECONDARY OUTCOMES:
Fatigue Severity Scale | At 6 and 12 months
  Clinical improvement
SAFTEE assessment | 1 month post last dose
  Adverse events
SF-36 continuous variables | 6 and 12 months
  Primary functional change with physical and mental summary indices as continuous variables.
SF-36 Responder-Nonresponder | 6 and 12 months
  Primary functional change with the physical and mental summary indices as either responder or nonresponder.
General Symptom Questionnaire | 6 and 12 months
  Changes in secondary clinical outcomes
PROMIS-29 | 6 and 12 months
  Changes in secondary clinical outcomes
Lyme VlsE1/pepC10 Antibody | 6 and 12 months
  Changes in quantitative antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher Paolino, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Upstate Global Health Institute, East Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies the primary results in a publication.
Time Frame: IPD will be shared with the primary publication.
Access Criteria: Primary IPD will be published with the primary manuscript describing the study. Requests for additional information can be requested by emailing warel@upstate.edu.